CLINICAL TRIAL: NCT02830295
Title: Physiotherapy in Mental Health: A Clinical Trial of Basic Body Awareness Therapy in Patients Suffering From Fibromyalgia
Brief Title: Effectiveness of Basic Body Awareness Therapy (BBAT) in Patients Suffering From Fibromyalgia
Acronym: BBAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cristina Bravo (Other)
Responsible Party: Sponsor-Investigator, Cristina Bravo, Principal investigator, Universitat de Lleida
Organization: Universitat de Lleida (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: University of Lleida
Record Dates: First submitted 2016-06-11; First posted 2016-07-12 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Fibromyalgia
Keywords: body awareness therapy; physical therapy; movement therapy
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Basic Body Awareness Therapy (Experimental): The Basic Body Awareness Therapy is usual therapy of physiotherapy in health mental in nord of europe. BBAT is based in twelve movements and massage that improve the movement quality of patient, also BBAT improves others movement qualities like biomechanical, physiologic, socio-cultural and existential.
  Interventions: Other: Basic Body Awareness Therapy
- control (No Intervention): the patients which below receive the treatment as usual, according the clinic guidelines of Health government

INTERVENTIONS:
Other: Basic Body Awareness Therapy — Basic body awareness therapy is a health oriented and person-centred approach with focus on the patient's resources. This is a method in physiotherapy, where we search to promote movement quality in daily life through self-exploration and self-experience.BBAT conceives the person from the biomechanical, physiological, bio-psycho-social and existential aspects, using the movement quality as a witness of the link in between all these perspectives.It can be done individually or in groups, through different daily life movements: lying, sitting, standing, walking, pair movements, use of voice and massages. BBAT has validated and reliable assesment tools, as BARS and BAS-I
  Other Names: BBAT (acronym)
  Arms: Basic Body Awareness Therapy

SUMMARY:
A randomized trial of Basic Body Awareness Therapy (BBAT) is applied in fibromyalgia patients as compared with a control intervention consisting of treatment as an usual. Sessions of BBAT lasted 90 minutes each and took place twice a week for 5 weeks. The primary end point is a change in the Visual Analog Scale score and Body Awareness Rating Scale and the secondary end points include Hospital Anxiety Depression, State Trait Anxiety Inventory, Beck Depression Inventory and Short Form 36. All assessments will be repeated at post treatment, 12 weeks and 24 weeks

DETAILED DESCRIPTION:
This work is a clinical trial of randomised and controlled groups. The hypothesis of study is that Basic Body Awareness Therapy applied in patients with fibromyalgia improves, more than usual treatment, the pain, normalization of postural pattern and movement, improve in psychologic state and improve of quality life.

The study population will be selected followed the inclusion criteria of fibromyalgia, and will be selected in area of primary health center, the patients will be divided in 2 groups, control group and treatment group. The groups will be examined at the begin, at 1 month of the begin of treatment, in 3 months, 6 months and one year to evaluated the outcomes in long time.

The dependence measurements will be Visual Analog Scale, Basic Body Awareness Rating Scale (BARS), SF-36, STAI A/R, BDI-II. The independence measurements will be demographic items: sex, age, country, level of studies, social status,..

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed of fibromyalgia according the American college of Rheumatology with 6 months at least
* the patients have to stay in different position as lying, sitting and standing

Exclusion Criteria:

* pregnancy
* suffering from another diseases that increase the pain or another specific diagnosis as rheumatic, heart disease and infectious disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-07; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | up to 24 weeks
  This scale evaluates the pain refered by patient with a scale from 0 to 10 being 10 the maximum pain

SECONDARY OUTCOMES:
Hospital Anxiety Depression | up to 24 weeks
  this scale evaluates the level of depression and anxiety with a questionary that score goes from 0 to 21, being 21 the maximum level of disease
Beck Depression Inventory | up to 24 weeks
  this scale evaluates the level of depression with a questionary that scores from 0 to 63, being 63 the maximum level of depression
State Trait Anxiety Inventory | up to 24 weeks
  this questionary evaluates the level of anxiety that scores from 0 to 60, being 60 the maximum level of anxiety
Short Form 36 | up to 24 weeks
  this questionary evaluates the quality of life in different components. The score goes from 0 to 100 being 100 the best score for quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Bravo Cristina, PT, Principal Investigator — Universitat de Lleida
Locations (1):
- Consorci Sanitari de l'Anoia, Igualada, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Gard G. Body awareness therapy for patients with fibromyalgia and chronic pain. Disabil Rehabil. 2005 Jun 17;27(12):725-8. doi: 10.1080/09638280400009071. PMID 16012065
- [Result] Courtois I, Cools F, Calsius J. Effectiveness of body awareness interventions in fibromyalgia and chronic fatigue syndrome: a systematic review and meta-analysis. J Bodyw Mov Ther. 2015 Jan;19(1):35-56. doi: 10.1016/j.jbmt.2014.04.003. Epub 2014 Apr 18. PMID 25603742
- [Result] Jones KD, King LA, Mist SD, Bennett RM, Horak FB. Postural control deficits in people with fibromyalgia: a pilot study. Arthritis Res Ther. 2011 Aug 2;13(4):R127. doi: 10.1186/ar3432. PMID 21810264